CLINICAL TRIAL: NCT00705315
Title: Docetaxel-epirubicin Plus Bevacizumab as First Line Therapy for Patients With Metastatic and HER2 Negative Breast Cancer. A Multicenter Phase I-II Study
Brief Title: Docetaxel/Epirubicin/Bevacizumab as First Line Therapy for Metastatic HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Dimitris Mavrudis, Hellenic Oncology Research Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/07.21
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; chemotherapy; biological therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Bevacizumab->Epirubicin->Docetaxel
  Interventions: Drug: Docetaxel; Drug: Epirubicin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel as an IV infusion over 1h at the dose of 75mg/m2 every 3 weeks for 6 cycles
  Other Names: Taxotere
Drug: Epirubicin — Epirubicin as an IV infusion over 10 min at the dose of 75mg/m2 every 3 weeks for 6 cycles
  Other Names: Farmorubicine
Drug: Bevacizumab — Bevacizumab as an IV infusion over 1h at the dose of 15 mg/kg every 3 weeks for 6 cycles
  Other Names: Avastin

SUMMARY:
This study will evaluate the efficacy and toxicity of docetaxel-epirubicin combination plus bevacizumab as first line treatment in patients with metastatic and HER2 negative breast cancer.

DETAILED DESCRIPTION:
A phase II trial with 142 patients demonstrated that therapy with docetaxel plus epirubicin is highly active first-line therapy for metastatic breast cancer, with acceptable toxicity profile. Recently initial therapy of metastatic breast cancer with paclitaxel plus bevacizumab demonstrated prolonged progression-free survival, as compared with paclitaxel alone. This study will evaluate the efficacy and toxicity of docetaxel-epirubicin combination plus bevacizumab as first line treatment in patients with metastatic and HER2 negative breast cancer. Furthermore, the efficacy of the combination therapy will be correlated with the presence of circulating tumor cells (CTCs) in this population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed metastatic breast adenocarcinoma
* No HER2 overexpression or gene amplification
* No previous therapy for metastatic breast cancer is allowed
* Age 18-75 years
* At least 12 months interval since prior adjuvant therapy with taxanes and/or anthracyclines
* Measurable disease as defined by the presence of at least one measurable lesion (except bone metastases, ascites or pleural effusions)
* Performance status (WHO) 0-2
* Adequate liver (serum bilirubin <1.5 times the upper normal limit, AST and ALT <2.5 times the upper normal limit in the absence of demonstrable liver metastases, or <5 times the UNL in the presence of liver metastases)
* Adequate renal function (serum creatinine <1.5 times the upper normal limit
* Adequate bone marrow function (neutrophils ≥ 1.5x 109 /L, and platelets ≥ 100x 109 /L)
* Written informed consent

Exclusion Criteria:

* Active infection
* Brain metastases
* History of significant cardiac disease (unstable angina, congestive heart failure, myocardial infarction within the previous 6 months, ventricular arrhythmias)
* History of stroke
* Anticoagulation therapy (except of low dose aspirin <325mg)
* Other invasive malignancy except nonmelanoma skin cancer
* Psychiatric illness or social situation that would preclude study compliance
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)

SECONDARY OUTCOMES:
Toxicity assessment | Toxicity assessment on each cycle
Time to Tumor Progression | 1 year
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Crete, Dep of Medical Oncology
Locations (10):
- Greece (10):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, 1st Dep of Medical Oncology, Athens
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - "Marika Iliadis" Hospital of Athens, Dep of Medical Oncology, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion
  - State General Hospital of Larissa, Dep of Medical Oncology, Larissa
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki

REFERENCES:
- [Derived] Tryfonidis K, Boukovinas I, Xenidis N, Christophyllakis C, Papakotoulas P, Politaki E, Malamos N, Polyzos A, Kakolyris S, Georgoulias V, Mavroudis D; Hellenic Oncology Research Group. A multicenter phase I-II study of docetaxel plus epirubicin plus bevacizumab as first-line treatment in women with HER2-negative metastatic breast cancer. Breast. 2013 Dec;22(6):1171-7. doi: 10.1016/j.breast.2013.08.017. Epub 2013 Oct 1. PMID 24091128